# **Statistical Analysis Plan**

LASARE: A Phase I Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses of 4P004 Versus Placebo Injected in the Target Knee Joint of Patients with Grade 2 to 4 Osteoarthritis on the Kellgren and Lawrence Severity Index.

Protocol Number: 4MB-LAS-P
Test Drug: Liraglutide
Sponsor: 4Moving Biotech
Date: 2023-11-27
Version: 1.0

Study LASARE - Statistical Analysis Plan v1.0 (2023-11-27) - CONFIDENTIAL

# **Names and Addresses**

The signatories agree to comply in all respects with this statistical analysis plan.

| | Name / Address |
|-----------------------------------------|----------------|
| SPONSOR | |
| Sponsor's legal representatives | |
| CLINICAL CRO | |
| CRO's legal representatives | |
| CDISC Packages and Statistical Analysis | |
| CRO's legal representatives | |

# Approvals

| Sponsor's Representative: | |
|---------------------------|----|
| Company: | |
| Signature: | |
| Date: | // |
| Artialis' representative: | |
| Signature: | |
| Date: | // |
| Statistician: | |
| Company: | |
| Signature: | |
| Date: | // |

# **Table of Contents**

| 1 | Abbreviations | 5 |
|-----|---------------------------------------------------------|----|
| 2 | Introduction | £ |
| | Purpose | |
| | Study Objectives | |
| | Study Design | |
| , | 5.1 Overall Study Design and Plan | |
| | 5.2 Method of Treatment Assignment and Randomization | |
| 6 | Sequence of Planned Analyses | 7 |
| | 6.1 Interim Analyses | 7 |
| | 6.2 Final Analyses and Reporting | 7 |
| 7 | Sample Size Estimation | 8 |
| 8 | Analysis Populations | 8 |
| 9 | General Principles for Statistical Analysis | 8 |
| | 9.1 Analysis Software | |
| | 9.2 Methods for Withdrawals, Missing Data, and Outliers | |
| | 9.3 Planned and Actual Treatment | |
| 4.0 | 9.4 Derived and Computed Variables | |
| 10 | Study Subjects | |
| | 10.2 Protocol Violations and Deviations | |
| 11 | Demographics and Other Baseline Characteristics | |
| 11 | 11.1 Demographics | |
| | 11.2 Prior Medications | |
| | 11.3 Medical History | |
| 12 | Safety and Tolerability Analyses | 10 |
| | 12.1 Concomitant Medications | 10 |
| | 12.2 Adverse Events | |
| | 12.2.1 Definitions | |
| | 12.2.2 Overview of TEAEs | |
| | 12.2.4 AESI | |
| | 12.2.5 Local tolerability | |
| | 12.2.6 Serious adverse events | |
| | 12.2.7 Deaths | |
| | 12.3 Target knee pain | |
| | 12.5 Vital Signs | |
| | 12.6 Electrocardiograms (ECG) | |
| | 12.7 Clinical safety laboratory assessment | |
| 13 | Pharmacokinetics Analyses | 17 |
| | 13.1 Endpoints | 17 |
| | 13.2 Plasma Concentration of Liraglutide | |
| | 13.3 Computation of PK Parameters | |
| | 13.4 Reporting of PK Parameters | |
| 14 | Exploratory Analyses | |
| 4- | 14.1 Endpoints | |
| 15 | Reporting Conventions | |
| | 15.1 General Reporting Conventions | |
| 16 | References | |
| | Tables, Figures & Listings in CSR Section 14 | |
| | Listings in CSR Section 16.2 | |
| 19 | Potentially Clinically Significant Abnormalities | 21 |

### 1 Abbreviations

AE Adverse event

AESI Adverse event of special interest ALT Alanine aminotransferase

AST Aspartate aminotransferase
ATC Anatomical therapeutic chemical

AUC Area under the curve
CrCl Creatinine clearance
Cmax Maximum concentration

CRF Case report form
CSR Clinical study report
DLT Dose Limiting toxicity

DSMB Data and safety monitoring board

ECG Electrocardiogram

eCRF Electronic case report form EMA European medical agency

EoS End of Study FU Follow up

GLP-1(R) Glucagon-like peptide 1 (receptor)

ICF Informed consent form

ICH International council for harmonisation

IA Intra-articular

IMP Investigational medicinal product KL Kellgren and Lawrence classification

MedDRA Medical dictionary for regulatory activities

MTD Maximum tolerated dose NRS Numerical rating scale

NSAID Nonsteroidal anti-inflammatory drug

OA Osteoarthritis

OARSI Osteoarthritis research society international PCSA Potentially clinically significant abnormality

PΚ Pharmacokinetic(s) PT Preferred term PTE Pre-treatment event SAE Serious adverse event SAP Statistical analysis plan SAS Statistical analysis system Standard deviation SD SOC System organ class

SUSAR Suspected unexpected serious adverse reaction

T1/2 Elimination half-life

TEAE Treatment-emergent adverse event

TK Target Knee

Tmax Time to maximum concentration

ULN Upper limit of normal

### 2 Introduction

This Statistical Analysis Plan (SAP) describes the planned analysis and reporting for clinical research study LASARE "A Phase I Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses of 4P004 Versus Placebo Injected in the Target Knee Joint of Patients with Grade 2 to 4 Osteoarthritis on the Kellgren and Lawrence Severity Index".

This study is being completed to characterize the safety and the tolerability of single IA administration of 4P004 at escalating doses (MTD) defined by occurrence of Dose Limiting Toxicities (DLTs).

The structure and content of this SAP provides sufficient detail to meet the requirements identified by the EMA and International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH): Guidance on Statistical Principles in Clinical Trials.

The following documents were reviewed in preparation of this SAP:

- Clinical Trial Protocol (4MB-LAS-P Version 3.0 July 2023)
- AdClin SOP "Clinical Data Analysis"
- ICH Guidance Topic E9 "Statistical Principles for Clinical Trials"
   [https://www.ema.europa.eu/en/documents/scientific-guideline/ich-e-9-statistical-principles-clinical-trials-step-5 en.pdf]

### 3 Purpose

The purpose of this SAP is to outline the planned analyses to be completed to support the completion of the Clinical Study Report (CSR) for the Clinical Trial Protocol 4MB-LAS-P, version 3.0 (17-07-2023), of the clinical research study LASARE "A Phase I Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses of 4P004 Versus Placebo Injected in the Target Knee Joint of Patients with Grade 2 to 4 Osteoarthritis on the Kellgren and Lawrence Severity Index". The planned analyses identified in this SAP will be included in regulatory submissions and/or future manuscripts.

Of note, since the study is primarily designed for safety and tolerability, complementary analyses may be performed to support the clinical development program. Any analysis performed but not identified in this SAP will be clearly identified in the respective CSR.

### 4 Study Objectives

The primary objectives are

- To characterize safety and tolerability of single IA administration of 4P004 at escalating doses
   in participants with knee OA grade 2 to 4 osteoarthritis (OA) on the Kellgren and Lawrence severity index (KL 2-4).
- To determine the maximum tolerated dose (MTD) defined by occurrence of Dose Limiting Toxicities (DLTs) in participants with knee OA KL 2-4.

The secondary objective is

 To characterize the plasma pharmacokinetics (PK) of liraglutide when administered as single IA doses at escalating dose levels in participants with knee OA KL 2-4.

The exploratory objective is

To collect biological fluids (blood, urine)

### 5 Study Design

### 5.1 Overall Study Design and Plan

Phase I study for IA injection, double-blind, placebo-controlled, randomized, multicenter, single ascending dose is designed to assess the safety, tolerability and pharmacokinetic of 4P004 in participants with target knee OA KL 2-4.

Participants were enrolled in 4 cohorts; in each cohort participants receive either 4P004 or placebo (6:2).

For the highest dose cohort, a sentinel dosing was planned and implemented.

Recruitment of participants

Participants are recruited via investigators' patient registry or via advertising.

- A Screening visit at D-7 (D-14 to D-4) is performed at study site and if the participant still agrees to participate in the study after the investigator has answered all his/her questions, the participant will sign the informed consent form.
   This visit should take place 4 to 14 days before the randomization day. During this visit, the eligibility of the participant will be evaluated.
- The Randomization visit (Day 1 to Day 2) is performed at study site and the participant is randomized in the study after review of inclusion & exclusion criteria. The participant will be hospitalized for 24 hours. The IMP IA injection will be performed by the investigator after a venous infusion line has been set up. Participant will be monitored during the 24-hour hospitalization and will be discharge on D2.
- The Follow-up visit at D4 (±1 day) is a virtual visit by phone call unless abnormal, clinically significant findings are observed upon discharge or at the investigator's discretion (participants should then be brought back to the clinic for re-evaluation).
- The Follow-up visit at D8 (±2 days) is a face-to-face visit. Participant will be asked to fill in a diary and a NRS questionnaire up to Day 29 to record any AE (in particular pain in the target knee) and analgesic medication taken.
- The End of Study (EoS) visit at D29 (±2 days) is a virtual visit by phone call unless abnormal, clinically significant findings are observed upon discharge or at the investigator's discretion (participants should then be brought back to the clinic for re-evaluation). Participant will be asked to send back to the Investigator the diary and the NRS questionnaire.

An independent Data and Safety Monitoring Board (DSMB) has been set up for this study and review safety data during the study. The DSMB is composed of 2 physicians specialized, one in rheumatology and one in diabetology. Members review the safety data in sessions on a regular basis during the study, and at any time if any SAE at least possibly related to liraglutide or safety issue occurs.

### 5.2 Method of Treatment Assignment and Randomization

Participants are enrolled in 4 cohorts; in each cohort participants receive either 4P004 or placebo (6:2).

Randomization has been performed using a pre-established randomization list. This list has been generated by a statistician for the IMPs (4P004 or placebo) based on study design (sequential randomization according to the dose escalation and sentinel patients).

The randomization is requested by the site at visit 2 (on D1) after eligibility confirmation. Participants are assigned their treatment according to the randomization schedule in the order in which they are randomized into the study.

### 6 Sequence of Planned Analyses

#### 6.1 Interim Analyses

No interim analysis is planned.

#### 6.2 Final Analyses and Reporting

All final, planned, analyses identified in the protocol and in this SAP will be performed only after the last patient has completed the study. A data review meeting will be held prior to database lock and completion of the final analyses.

In addition, no database may be locked, or analyses completed until this SAP has been approved.

Key statistics and study results will be made available following database lock and prior to completion of the final clinical study report (CSR).

Any, post-hoc, exploratory analyses completed to support planned study analyses, which are not identified in this SAP, will be documented and reported in appendices to the CSR. Any results from these unplanned analyses will also be clearly identified in the text of the CSR.

### 7 Sample Size Estimation

The sample size was not based on statistical power considerations. The sample size for this study of 8 participants in each cohort (6 active : 2 placebo) is considered to be sufficient for evaluation of safety, tolerability, and PK of each cohort.

### 8 Analysis Populations

The following analysis populations are defined for the study:

- Safety population: The safety analysis set will consist of all participants who are enrolled and received 1 dose of study drug.
- PK population: The Pharmacokinetics (PK) analysis set will consist of all participants who receive study drug and have at least 1 measurable plasma concentration. Placebo subjects will not be part of the PK population.

Unless otherwise stated, all analyses will be done on the Safety population.

### 9 General Principles for Statistical Analysis

Data will be summarized using classical descriptive statistics for the following groups:

- pooled placebo (i.e. participants receiving placebo in any cohort),
- each 4P004 dose level,
- unplanned doses if any (see below),
- 4P004 overall

A group "All" (Placebo + 4P004 overall) will be added if explicitly mentioned.

Categorical data will be presented using counts and percentages of subjects, while continuous variables will be presented using the mean, standard deviation, median, minimum, maximum, and number of observations with non-missing values. The coefficient of variation [%CV] will be provided for PK parameters.

The safety evaluation will be based upon the review of the individual values and descriptive statistics. No statistical significance tests will be performed on safety data.

### 9.1 Analysis Software

Statistical analysis will be performed using SAS version 9.4 for Windows or later.

### 9.2 Methods for Withdrawals, Missing Data, and Outliers

Missing data will not be replaced. Analyses will be done on the maximum available observed data. If a PK point is missing at time t, an interpolation may be done, depending on data review.

#### 9.3 Planned and Actual Treatment

In cohort 3 one participant was underdosed; the Sponsor decided (blinded review) to include one more participant to ensure 6 participants with the right active dose; consequently a ninth participant has been included to receive the same treatment as the underdosed participant. Therefore, at least one subject may have an actual treatment different from the planned one (if the underdosed subject did not receive placebo).

Participants who did not receive the planned treatment will be assigned, upon review of their actual treatment, to either of the following actual arm:

if the received treatment is one of the planned ones, or close enough, to the corresponding arm

otherwise, to an arm "4P004 unplanned"

Unless stated otherwise, analyses will be presented by actual arm.

### 9.4 Derived and Computed Variables

For any variable, the baseline value is defined as the last observation before IMP injection.

The time will be split into 3 periods (epochs):

- before treatment (screening)
- during treatment (from IMP injection to 7 days after IMP injection date)

after treatment

The following PK parameters will be calculated from measured plasma concentrations for each participant:

- Maximum observed concentration (Cmax)
- Time of maximum observed concentration (Tmax)
- Area under the curve (AUC<sub>0-t</sub>)
- Terminal Half-life (T<sub>1/2</sub>)

### 10 Study Subjects

### 10.1 Disposition of Participants and Withdrawals

**Table TTT. Participant disposition** 

| | Placebo | 4P004 | 4P004 | 4P004 | 4P004 | 4P004 | All |
|---|---|---|---|---|---|---|---|
| | (pooled) | | | | | (pooled) | |
| Screened Participants | | | | | | | XX |
| Randomized Subjects <sup>1</sup> | XX | XX | XX | XX | XX | XX | XX |
| Treated Subjects <sup>2</sup> | XX | XX | XX | XX | XX | XX | XX |
| Completed Subjects <sup>2</sup> | XX | XX | XX | XX | XX | XX | XX |
| Withdrawn Subjects <sup>2</sup> | XX | XX | XX | XX | XX | XX | XX |
| Reason 1 | XX | XX | XX | XX | XX | XX | XX |
| ••• | XX | XX | XX | XX | XX | XX | XX |

<sup>&</sup>lt;sup>1</sup> by planned treatment

#### 10.2 Protocol Violations and Deviations

Protocol violations and deviations are not described in the protocol, and will be established by blind review.

Major deviations are defined as follows:

- non respect of inclusion criteria
- underdose
- overdose

All others will be considered as minor deviations.

### **Table TTT. Deviations by Category**

Major, Minor

Major deviations will be listed:

#### **Listing LLL. Major Deviations**

Subject Id, Treatment Group, Deviation Text

### 11 Demographics and Other Baseline Characteristics

All TFL in this section will include the column "All".

#### 11.1 Demographics

#### **Table TTT. Demographics and Baseline Characteristics**

Sex, Age, Weight, BMI, KL Grade, Pain at Visit 2 (mean of the previous 48h)

#### **Table TTT. Other Baseline Characteristics**

Height, Race

#### 11.2 Prior Medications

Medication will be coded using the WHO-ATC/DDD Index 2023.

All tables in this section will be sorted by descending percentages in the column "4P004 (pooled)".

Medications will be flagged with 3 flags:

pre-treatment: treatment taken during screening

<sup>&</sup>lt;sup>2</sup> by actual treatment

- on-treatment: treatment taken during the treatment period
- post-treatment: treatment taken after the treatment period

In case of uncertainty, a medication will be assigned to all periods during which it might have been taken.

Medications not classified as pain killer vs. other medications will be assigned to one of the two categories for analyses, based on medical review by the Sponsor

Table TTT. Pain killers started and ended before treatment

| ATC Level 2 | Placebo | 4P004 | 4P004 | 4P004 | 4P004 | 4P004 | All |
|---|---|---|---|---|---|---|---|
| | (pooled) | | | | | (pooled) | |
| | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Any pain killer | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC 2 term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC 2 term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Table TTT. Other medications started and ended before treatment

| ATC Level 2 | Placebo | 4P004 | 4P004 | 4P004 | 4P004 | 4P004 | All |
|---|---|---|---|---|---|---|---|
| | (pooled) | | | | | (pooled) | |
| | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Any medication | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC 2 term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC 2 term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

### 11.3 Medical History

All tables in this section will be sorted by descending percentages in the column "4P004 (pooled)".

**Table TTT. Medical History by SOC** 

| SOC | Placebo | 4P004 | 4P004 | 4P004 | 4P004 | 4P004 | All |
|---|---|---|---|---|---|---|---|
| | (pooled) | | | | | (pooled) | |
| | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Any Medical History | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| SOC term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| SOC term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

## 12 Safety and Tolerability Analyses

#### 12.1 Concomitant Medications

All tables in this section will be sorted by descending percentages in the column "4P004 (pooled)".

Table TTT. Pain killers started before treatment and continuing at IMP injection

| ATC Level 2 | Placebo | 4P004 | 4P004 | 4P004 | 4P004 | 4P004 | All |
|---|---|---|---|---|---|---|---|
| | (pooled) | | | | | (pooled) | |
| | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Any pain killer | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC 2 term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC 2 term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC 4 term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| () | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Table TTT. Other medications started before treatment and continuing at IMP injection

| ATC Level 2 | Placebo | 4P004 | 4P004 | 4P004 | 4P004 | 4P004 | All |
|---|---|---|---|---|---|---|---|
| ATC Level 4 | (pooled) | | | | | (pooled) | |
| | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Any medication | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC 2 term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC 4 term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| () | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC 2 term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC 4 term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| () | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Table TTT. Pain killers started during treatment

| ATC Level 2 | Placebo | 4P004 | 4P004 | 4P004 | 4P004 | 4P004 |
|---|---|---|---|---|---|---|
| ATC Level 4 | (pooled) | | | | | (pooled) |
| | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Any pain killer | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

| ATC 2 term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
|---|---|---|---|---|---|---|
| ATC 4 term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| () | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC 2 term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC 4 term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| () | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Table TTT. Other medications started during treatment

| ATC Level 2 | Placebo | 4P004 | 4P004 | 4P004 | 4P004 | 4P004 |
|---|---|---|---|---|---|---|
| ATC Level 4 | (pooled) | | | | | (pooled) |
| | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Any medication | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC 2 term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC 4 term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| () | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC 2 term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC 4 term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| () | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

### 12.2 Adverse Events

All tables in this section will be sorted by descending percentages in the column "4P004 (pooled)".

#### 12.2.1 Definitions

Adverse events will be classified in one of three categories:

- pre-treament: events that certainly started during screening
- post-treatment: events that certainly started after the treatment period
- treatment-emergent (TEAE): all other events

#### 12.2.2 Overview of TEAEs

This table will also show the number of AEs, as depicted below.

**Table TTT. Overview of TEAEs** 

| | Placebo | | 4P004 | | 4P004 | | 4P004 | | 4P004 | | 4P004 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (pooled) | | | | | | | | | | (pooled) | |
| | (N=XX) | | (N=XX) | | (N=XX) | | (N=XX) | | (N=XX) | | (N=XX) | |
| | Subjects | # <sup>1</sup> | Subjects | # <sup>1</sup> | Subjects | # <sup>1</sup> | Subjects | # <sup>1</sup> | Subjects | # <sup>1</sup> | Subjects | #1 |
| Any TEAE | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX |
| AESI | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX |
| SAEs | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX |
| by Toxicity Grade | | | | | | | | | | | | |
| 1 Mild | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX |
| 2 Moderate | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX |
| by Relationship to Study Drug | | | | | | | | | | | | |
| Not Related | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX |
| Unlikely | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX |
| () | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX |
| by Outcome | | | | | | | | | | | | |
| Recovered | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX |
| Recovering | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX |
| () | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX | XX (X.X%) | XX |

<sup>&</sup>lt;sup>1</sup> Numbers of adverse events

### 12.2.3 All TEAEs

Table TTT. TEAEs by SOC and PT

| SOC | Placebo | 4P004 | 4P004 | 4P004 | 4P004 | 4P004 |
|---|---|---|---|---|---|---|
| PT | (pooled) | | | | | (pooled) |
| | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Any TEAE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| SOC term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| PT term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| () | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| SOC term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| PT term | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| () | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Table TTT. TEAEs by SOC, PT and Toxicity Grade

| SOC | Toxicity | Placebo | 4P004 | 4P004 | 4P004 | 4P004 | 4P004 |
|---|---|---|---|---|---|---|---|
| PT | Grade | (pooled) | | | | | (pooled) |
| | | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Any TEAE | 1 Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 2 Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | () | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| SOC term | 1 Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 2 Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | () | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| PT term | 1 Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 2 Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | () | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| () | | | | | | | |
| SOC term | 1 Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 2 Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | () | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| PT term | 1 Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 2 Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | () | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| () | | • | • | • | • | • | |

With the same template, the TEAEs will be presented by Relationship to study drug, grouped as:

- Not related: No/Unlikely
- Related: Possible, Probable, Definite

#### Table TTT. TEAEs by SOC, PT and Relationship to Study Drug

#### 12.2.4 AESI

AESI defined in the protocol are:

- Pregnancy of the participant or of his partner
- Symptomatic overdose
- Anaphylaxis
- Severe IMP injection site reactions
- Hypoglycemia
- Severe gastro-intestinal disorder

All tables in the section "All TEAEs" will be reproduced for TEAEs of SI, except by relationship to study drug. All tables will also show the number of adverse events, as in the Overview of Adverse Events.

#### Table TTT. Treatment-Emergent AESIs by SOC and PT

### Table TTT. Treatment-Emergent AESIs by SOC, PT and Toxicity Grade

A listing of all treatment-emergent AESI will also be provided.

### **Listing LLL. Treatment-Emergent AESIs**

#### 12.2.5 Local tolerability

The AE details in case of severe IMP injection site reaction will be presented as follows:

**Table TTT. Injection Site Reactions** 

| Kind of | Maximum | Placebo | 4P004 | 4P004 | 4P004 | 4P004 | 4P004 |
|---|---|---|---|---|---|---|---|
| Reaction | Toxicity | (pooled) | | | | | (pooled) |
| | Grade | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Any Kind | Any Grade | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 1 Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 2 Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | () | | | | | | |
| Tenderness | Any Grade | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 1 Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 2 Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | () | | | | | | |
| Erythema | Any Grade | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 1 Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 2 Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | () | | | | | | |
| () | • • | | | | | | |

#### 12.2.6 Serious adverse events

A listing of all SAEs will be provided.

#### **Listing LLL. Serious Adverse Events**

#### 12.2.7 Deaths

If any subject dies during the study, relevant information will be supplied in a data listing, and appropriate SAE narratives.

#### **Listing LLL. Deaths**

#### 12.3 Target knee pain

The target knee pain, evaluated on a 0-10 scale, is measured as follows:

| Visit | Timepoint | Table |
|--------------|-------------------------------------------|-------|
| Screening | (mean of the last 48 hours) | - |
| Visit 2 | (mean of the last 48 hours) | 2,3 |
| | Pre-Dose | 1 |
| | 1h Post-Dose | 1 |
| | 2h Post-Dose | 1 |
| | 3h Post-Dose | 1 |
| | 4h Post-Dose | 1 |
| | 5h Post-Dose | 1 |
| | 6h Post-Dose | 1 |
| | 24h Post-Dose (mean of the last 24 hours) | 1,2,3 |
| Visit 3 | (mean of the last 24 hours) | 2,3 |
| | Day 3 (mean of the last 24 hours) | 3 |
| | Day 4 (mean of the last 24 hours) | 3 |
| | Day 5 (mean of the last 24 hours) | 3 |
| | Day 6 (mean of the last 24 hours) | 3 |
| | Day 7 (mean of the last 24 hours) | 3 |
| | Day 8 (mean of the last 24 hours) | 3 |
| Phone Call 2 | Day 15 (mean of last 48 hours) | 2 |
| | Day 22 (mean of last 48 hours) | 2 |
| | Day 29 (mean of last 48 hours) | 2 |

In the tables of this section, in addition to the values, the change from Baseline will be added, with the standard summary statistics and the number of subjects with an aggravation since the Baseline.

In case of two different measures on the same day, the value of the diary will prevail.

The pain will be presented in three summary tables:

#### Table TTT. Target Knee Pain from Pre-Dose to 24h Post-Dose

(timepoints marked « table 1 » in the list above)

#### Table TTT. Target Knee Pain from Visit 2 to End of Study

(timepoints marked « table 2 » in the list above)

For this table, the baseline will be the mean of the last 48 hours collected at Visit 2 or, if not available, the Screening value.

#### Table TTT. Target Knee Pain from Visit 2 to Day 8

(timepoints marked « table 3 » in the list above)

This table will be presented by actual day of pain, whatever scheduled day the measure has been assigned to.

#### 12.4 Weight

Weight will be presented at Baseline and at Visit 3, with the change from Baseline.

#### **Table TTT. Weight over Time**

#### 12.5 Vital Signs

The vital signs are systolic blood pressure, diastolic blood pressure and heart rate. They are measured as follows:

| Visit | Timepoint |
|-----------|---------------|
| Screening | - |
| Visit 2 | Pre-Dose |
| | 1h Post-Dose |
| | 2h Post-Dose |
| | 4h Post-Dose |
| | 8h Post-Dose |
| | 12h Post-Dose |
| | 24h Post-Dose |
| Visit 3 | _ |

The following will be presented for each vital sign:

- value (mean, SD, etc.)
- absolute change from baseline (mean, SD, etc.)
- PCSA (frequencies and percentages)

**Table TTT. Systolic Blood Pressure over Time** 

| mmHg | Placebo | 4P004 | 4P004 | 4P004 | 4P004 | 4P004 |
|---|---|---|---|---|---|---|
| | (pooled) | | | | | (pooled) |
| | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Baseline | | | | | | |
| Value | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| mean (SD) | XX (XX) | XX (XX) | XX (XX) | XX (XX) | XX (XX) | XX (XX) |
| () | | | | | | |
| 1h Post-Dose | | | | | | |
| Value | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| mean (SD) | XX (XX) | XX (XX) | XX (XX) | XX (XX) | XX (XX) | XX (XX) |
| () | | | | | | |
| Change from BL | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| mean (SD) | XX (XX) | XX (XX) | XX (XX) | XX (XX) | XX (XX) | XX (XX) |
| () | | | | | | |
| PCSA | | | | | | |
| ≤ 95 + decrease from baseline ≥ 20 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ≥ 160 + increase from baseline ≥ 20 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| No PCSA | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| () | | | | | | |

#### **Table TTT. Heart Rate Pressure over Time**

### 12.6 Electrocardiograms (ECG)

The 12-lead ECG parameters are Heart Rate, PR, QRS and QT. They are measured at the following times: Screening (D-7), D1 (T0-15min and T0+12h).

They will be presented with the same layout as Vital Signs, at Baseline and 12 hours post-baseline. The relative change from baseline will be added.

Table TTT. ECG: Hear Rate over Time

Table TTT. ECG: PR over Time

Table TTT. ECG: QRS over Time

Table TTT. ECG: QT over Time

### 12.7 Clinical safety laboratory assessment

The Hematology and Chemistry parameters are collected at Screening and Visit 3.

They are:

#### Hematology:

- Erythrocytes
- Hemoglobin
- Hematocrit
- Leukocytes
- Monocytes
- Neutrophils
- $\ \ Eosinophils$
- Basophils
- LymphocytesPlatelets

### Chemistry:

- Creatinine Clearance
- Potassium
- Chloride
- Sodium
- Calcium
- Alanine Aminotransferase
- Aspartate Aminotransferase
- Amylase
- Glucose (at Screening and Visit 3)

They will be presented like Vital Signs, but with one table for Hematology, one for Chemistry.

**Table TTT. Hematology over Time** 

| | Placebo | 4P004 | 4P004 | 4P004 | 4P004 | 4P004 |
|---|---|---|---|---|---|---|
| | (pooled) | | | | | (pooled) |
| | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Erythrocytes (tera/L) | | | | | | |
| Baseline | | | | | | |
| Value | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| mean (SD) | XX (XX) | XX (XX) | XX (XX) | XX (XX) | XX (XX) | XX (XX) |
| () | | | | | | |
| PCSA | | | | | | |
| ≤ 95 + decrease from baseline ≥ 20 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ≥ 160 + increase from baseline ≥ 20 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| No PCSA | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Visit 3 | | | | | | |
| Value | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| mean (SD) | XX (XX) | XX (XX) | XX (XX) | XX (XX) | XX (XX) | XX (XX) |
| () | | | | | | |
| Change from BL | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| mean (SD) | XX (XX) | XX (XX) | XX (XX) | XX (XX) | XX (XX) | XX (XX) |
| () | | | | | | |
| PCSA | | | | | | |
| ≤ 95 + decrease from baseline ≥ 20 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ≥ 160 + increase from baseline ≥ 20 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| No PCSA | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| () | | | | | | |

For parameters with defined PCSA, a table with PCSA only will be produced:

**Table TTT. Hematology PCSA over Time** 

| | Placebo | 4P004 | 4P004 | 4P004 | 4P004 | 4P004 |
|---|---|---|---|---|---|---|
| | (pooled) | | | | | (pooled) |
| | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Erythrocytes (tera/L) | | | | | | |
| Baseline | | | | | | |
| ≤ 95 + decrease from baseline ≥ 20 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ≥ 160 + increase from baseline ≥ 20 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| No PCSA | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Visit 3 | | | | | | |
| ≤ 95 + decrease from baseline ≥ 20 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ≥ 160 + increase from baseline ≥ 20 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| No PCSA | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| () | | | | | | |

### **Table TTT. Chemistry over Time**

### **Table TTT. Chemistry PCSA over Time**

Glycemia is measured as follows:

| Visit | Timepoint | Method |
|-----------|---------------|--------------------|
| Screening | - | Blood |
| Visit 2 | Pre-Dose | Blood & Glucometer |
| Visit 2 | 1h Post-Dose | Glucometer |
| Visit 2 | 2h Post-Dose | Blood |
| Visit 2 | 4h Post-Dose | Blood |
| Visit 2 | 6h Post-Dose | Glucometer |
| Visit 2 | 8h Post-Dose | Blood |
| Visit 2 | 10h Post-Dose | Glucometer |
| Visit 2 | 12h Post-Dose | Blood |
| Visit 2 | 16h Post-Dose | Blood |
| Visit 2 | 24h Post-Dose | Glucometer |
| Visit 3 | - | Blood & Glucometer |

In order to obtain one value per scheduled timepoint:

- The baseline value will be selected as the last measure before IMP injection. If there are such two measures (same time, different method), then Blood will be selected.
- Post-baseline, if there are two measures for a scheduled timepoint, Blood will be selected.
- Additional samples vs. scheduled samples will not be analyzed, unless they are the baseline.

The values will be reported over time (Baseline, 1h Post-Dose to 24h Post-Dose) with the same template as Vital Signs.

#### Table TTT. Glycemia over Time

### 13 Pharmacokinetics Analyses

Pharmacokinetics analysis will be done on the PK population.

Blood samples for placebo will not be analyzed by the bioanalytical laboratory except for 2 samples per participant receiving placebo, 1 pre-dose and the other at 12h post-dose, to confirm that these participants did not receive liraglutide. These results will be listed in section 16.2 of the CSR.

The placebo group will not be presented in the TFL of this section. In summary tables, only the columns corresponding to the doses will be presented (no "pooled" column).

In this section only, the treatment groups will show the real dose administered, in case the real dose is not one of the scheduled ones.

#### 13.1 Endpoints

The endpoints are:

- Plasma concentration of Liraglutide following a single IA injection at D1 (pre-injection T0-15 min), and 2, 4, 8, 12, 16 and 24 hours post-injection.
- The PK parameters Cmax, Tmax, AUC0-t and T1/2.

#### 13.2 Plasma Concentration of Liraglutide

A summary table will be produced by timepoint:

#### Table TTT. Plasma Concentrations over Time

The plasma concentrations over time will be plotted for each subject, on both arithmetic and logarithmic scales. There will be one series of figures for all subjects at a given dose.

Figure FFF. Plasma Concentrations over Time by Subject - Dose



Figure FFF. Plasma Concentrations over Time by Subject - Dose



Figure FFF. Plasma Concentrations over Time by Subject - Dose



Figure FFF. Plasma Concentrations over Time by Subject - Dose

#### 13.3 Computation of PK Parameters

In case of missing concentration, the individual figure of PK concentrations of the subject will be reviewed, and a decision will be made:

- interpolate the concentration or not
- possibly invalidate some PK parameters (set them to missing)

Concentrations BLOQ will be set to zero if measured at baseline, to LLOQ/2 otherwise.

The parameters will be derived as follows:

- Cmax Maximum concentration achieved computed as max(C0-C6)
- Tmax Time to reach maximum concentration computed as first time Ti where Concentration = Cmax

- AUC0-t The area under the concentration vs. Time curve computed as follows:
  - Tlast = last time where Clast > BLOQ
  - AUC0-t = sum of AUCs using linear trapezoidal summation from time 0 to Tlast
- λz terminal elimination rate constant

computed as follows:

- select the timepoints t1 = T0+16h and t2 = T0+24h, with respective concentrations C1 and C2
- if either concentration is missing,  $\lambda z$  is missing
- otherwise, compute the slope of the line ln(C1) to ln(C2)
- if the slope is negative,  $\lambda z = -slope$
- otherwise λz is missing
- $T1/2 = In(2) / \lambda z$

The dose-normalized parameters Cmax and AUCO-t will also be computed (Cmax/Dose and AUCO-t/Dose).

### 13.4 Reporting of PK Parameters

The PK parameters will be summarized. In addition to standard univariate statistics, the coefficient of variation, geometric mean and geometric standard deviation will be added.

**Table TTT. PK Parameters** 

### 14 Exploratory Analyses

Exploratory analysis will be done on the Safety set.

#### 14.1 Endpoints

The endpoints are:

Serum and urine OA-related biomarkers (exploratory proteomic research of 4P004 efficacy related biomarkers) at D1 (T0-15min, 8h, 24h) and D8.

The exploratory endpoint will be analyzed separately, and the related data will not be included in the SDTM/ADaM datasets.

### 15 Reporting Conventions

The following reporting conventions will be adopted for the SAP. These conventions will enhance the review process and help to standardize presentation with common notations.

### 15.1 General Reporting Conventions

Legends will be used for figures with more than one variable or item displayed.

All date values will be presented as YYYY-MM-DD (e.g., 2001-08-29) format.

As a general rule, percentages will be presented with one decimal digit, but can be presented with no decimal digit for table width requirements.

#### **15.2 Population Summary Conventions**

The biomarker concentration in serum determined at each sampling time point should be presented on the original scale for each subject participating in the study.

Population(s) identified in all TFL titles as "All Subjects", "Safety Population" or "PK Population".

#### 16 References

ICH Guidance Topic E9 "Statistical Principles for Clinical Trials"

# 17 Tables, Figures & Listings in CSR Section 14

The following tables will be included in the report either in the text or in a dedicated chapter reporting all tables but not included in the text.

| Туре | Number | Title | Population |
|---|---|---|---|
| Table | 1.1 | Participant disposition | All |
| Table | 1.2 | Deviations by Category | Safety |
| Listing | 1.2.1 | Major Deviations | Safety |
| Table | 1.3 | Demographics and Baseline Characteristics | Safety |
| Table | 1.4 | Other Baseline Characteristics | Safety |
| Table | 1.5.1 | Pain killers started and ended before treatment | Safety |
| Table | 1.5.2 | Other medications started and ended before treatment | Safety |
| Table | 1.6 | Medical History by SOC | Safety |
| Table | 2.1 | Pain killers started before treatment and continuing at IMP injection | Safety |
| Table | 2.2 | Pain killers started during treatment | Safety |
| Table | 2.3 | Other medications started before treatment and continuing at IMP injection | Safety |
| Table | 2.4 | Other medications during treatment | Safety |
| Table | 3.1 | Overview of TEAEs | Safety |
| Table | 3.1.1 | TEAEs by SOC and PT | Safety |
| Table | 3.1.2 | TEAEs by SOC, PT and Toxicity Grade | Safety |
| Table | 3.1.3 | TEAEs by SOC, PT and Relationship to Study Drug | Safety |
| Table | 3.2 | Treatment-Emergent AESIs by SOC and PT | Safety |
| Table | 3.2.1 | Treatment-Emergent AESIs by SOC, PT and Toxicity Grade | Safety |
| Listing | 3.2.2 | Treatment-Emergent AESIs | Safety |
| Table | 3.3 | Injection Site Reactions | Safety |
| Listing | 3.4 | Serious Adverse Events | Safety |
| Listing | 3.5 | Deaths | Safety |
| Table | 4.1 | Target Knee Pain from Pre-Dose to 24h Post-Dose | Safety |
| Table | 4.2 | Target Knee Pain from Visit 2 to End of Study | Safety |
| Table | 4.3 | Target Knee Pain from Visit 2 to Day 8 | Safety |
| Table | 5.0 | Weight over Time | Safety |
| Table | 5.1 | Systolic Blood Pressure over Time | Safety |
| Table | 5.2 | Diastolic Blood Pressure over Time | Safety |
| Table | 5.3 | Heart Rate over Time | Safety |
| Table | 6.1 | ECG: Heart Rate over Time | Safety |
| Table | 6.2 | ECG: PR over Time | Safety |
| Table | 6.3 | ECG: QRS over Time | Safety |
| Table | 6.4 | ECG: QT over Time | Safety |
| Table | 7.1 | Hematology over Time | Safety |
| Table | 7.1.1 | Hematology PCSA over Time | Safety |
| Table | 7.2 | Chemistry over Time | Safety |
| Table | 7.2.1 | Chemistry PCSA over Time | Safety |
| Table | 7.3 | Glycemia over Time | Safety |
| Table | 8.1 | Plasma Concentrations over Time | PK |
| Figure | 8.1.0.3 | Plasma Concentrations over Time by Subject - | PK |
| Figure | 8.1.1 | Plasma Concentrations over Time by Subject - | PK |
| Figure | 8.1.2 | Plasma Concentrations over Time by Subject - | PK |
| Figure | 8.1.3 | Plasma Concentrations over Time by Subject - | PK |
| Table | 8.2 | PK Parameters | PK |

# 18 Listings in CSR Section 16.2

The following listings will be included in section 16.2 of the CSR.

| Type | Number | Title | Population |
|---------|---------|----------------------------------------|------------|
| Listing | 16.2.1 | Demographics and Disposition | Safety |
| Listing | 16.2.2 | Prior and Concomitant Medications | Safety |
| Listing | 16.2.3 | Medical History | Safety |
| Listing | 16.2.4 | Serology | Safety |
| Listing | 16.2.5 | Knee X-Ray and Kellgren-Lawrence Grade | Safety |
| Listing | 16.2.6 | Failed Inclusion/Exclusion Criteria | Safety |
| Listing | 16.2.7 | IMP Injection | Safety |
| Listing | 16.2.8 | Deviations | Safety |
| Listing | 16.2.9 | Adverse Events | Safety |
| Listing | 16.2.10 | Knee Pain Assessments | Safety |
| Listing | 16.2.11 | Height, Weight and BMI | Safety |
| Listing | 16.2.12 | Vital Signs | Safety |
| Listing | 16.2.13 | ECG | Safety |
| Listing | 16.2.14 | Hematology | Safety |
| Listing | 16.2.15 | Chemistry | Safety |
| Listing | 16.2.16 | Glycemia | Safety |
| Listing | 16.2.17 | Exploratory Sample Collection | Safety |
| Listing | 16.2.18 | Plasma Concentrations | Safety |
| Listing | 16.2.19 | PK Parameters | Safety |
| Listing | 16.2.20 | Visits | Safety |

# 19 Potentially Clinically Significant Abnormalities

Potentially clinically significant abnormality (PCSA) values are defined as abnormal values considered medically important by the Sponsor, according to predefined criteria/thresholds based on literature reviews and defined by the Sponsor for clinical laboratory tests, vital signs, and ECG parameters.

When possible, PCSA will be computed at baseline or before.

| Parameter | PCSA | Comments |
|---|---|---|
| Chemistry | | |
| AST or ALT | > 3 ULN | Guidance for Industry Drug-Induced Liver Injury FDA, 2009 |
| Potassium | < 3 mmol/L or ≥ 5.5 mmol/L | |
| CLcr (mL/min)<br>(Estimated creatinine<br>clearance based on<br>the Cokcroft Gault<br>equation) | < 15 (end stage renal disease) ≥ 15 - < 30 (severe decrease in GFR) ≥ 30 - < 60 (moderate decrease in GFR) | FDA draft Guidance 2020 Pharmacokinetics in Patients with Impaired Renal Function Study Design, Data Analysis, and Impact on Dosing |
| Amylasemia | ≥ 1.5 ULN | |
| Glycemia | < 70 mg/dL | DSMB |
| Hematology | | |
| RBC | ≥ 6 Tera/L | |
| Hb | ≤ 115 g/L (Male); ≤ 95 g/L (Female)<br>≥ 185 g/L (Male); ≥ 165 g/L (Female)<br>Decrease from Baseline ≥ 20 g/L | Criteria based upon decrease from baseline are more relevant than based on absolute value. |
| WBC | < 3.0 Giga/L (Non-Black)<br>< 2.0 Giga/L (Black)<br>≥ 16.0 Giga/L | |
| Lymphocytes | > 4.0 Giga/L | |
| Neutrophils | < 1.5 Giga/L (Non-Black);<br>< 1.0 Giga/L (Black) | International Consensus meeting on drug-<br>induced blood cytopenias, 1991.<br>FDA criteria. |
| Monocytes | > 0.7 Giga/L | |
| Basophils | > 0.1 Giga/L | |
| Eosinophils | > 0.5 Giga/L | Harrison- Principles of internal Medicine 17th Ed., 2008 |
| Platelets | < 100 Giga/L<br>≥ 700 Giga/L | International Consensus meeting on drug-<br>induced blood cytopenias, 1991. |
| Vital Signs | | |
| HR (bpm) | ≤ 50 + decrease from baseline ≥ 20<br>≥ 120 + increase from baseline ≥ 20 | |
| SBP (mmHg) | ≤ 95 + decrease from baseline ≥ 20<br>≥ 160 + increase from baseline ≥ 20 | |
| DBP (mmHg) | ≤ 45 + decrease from baseline ≥ 10<br>≥ 110 + increase from baseline ≥ 10 | |
| ECG | | |
| HR (bpm) | < 50<br>< 50 + decrease from baseline ≥ 20<br>> 100<br>> 100 + increase from baseline ≥ 20 | |
| PR (ms) | > 200<br>> 200 + increase from baseline ≥ 25% | |
| QRS (ms) | > 110<br>> 110 + increase from baseline ≥ 25% | |
| QT (ms) | > 500 | |